CLINICAL TRIAL: NCT00818220
Title: Protective Effects of Delayed Cord Clamping in VLBW Infants
Brief Title: Protective Effects of Delayed Cord Clamping in Very Low Birth Weight (VLBW) Infants
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Rhode Island (Other)
Collaborators: Women and Infants Hospital of Rhode Island (Other); Brown University (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Judith S Mercer, Clinical Professor, University of Rhode Island
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2980022; 5R01NR010015-02 (NIH)
Record Dates: First submitted 2009-01-05; First posted 2009-01-07 (Estimated); Last update posted 2015-05-27 (Estimated); Status verified 2015-05

CONDITIONS: Intraventricular Hemorrhage; Sepsis
Keywords: intraventricular hemorrhage; sepsis; motor function; motor functioning at 7 months corrected age; cytokines in cord blood and at 6 and 20 hours of age; stem cells in cord blood and at 20 hours of age
MeSH Terms: conditions — Sepsis | interventions — Umbilical Cord Clamping

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1-Delayed Cord Clamping (DCC) (Experimental): Immediately after birth, the infant is placed in a warm blanket and held lower than the placenta. The research nurse counts out 30 to 45 seconds for the obstetrician. The cord is milked once and then clamped at 30 to 45 seconds after birth.
  Interventions: Procedure: delayed umbilical cord clamping
- 2-Immediate Cord Clamping (ICC) (Active Comparator): Routine care which is immediate cord clamping
  Interventions: Other: Immediate cord clamping

INTERVENTIONS:
Procedure: delayed umbilical cord clamping — at birth, the clamping of the umbilical cord will be delayed 30 to 45 seconds while the child is held lower than the placenta. At the end of the time, the cord is milked once and the cord is clamped. If the obstetrician feels he cannot delay the cord clamping, then the cord can be milked 2 to 3 times.
  Other Names: immediate cord clamping; cord milking
  Arms: 1-Delayed Cord Clamping (DCC)
Other: Immediate cord clamping — The umbilical cord is cut within 10 seconds after birth
  Other Names: routine care
  Arms: 2-Immediate Cord Clamping (ICC)

SUMMARY:
The purpose of this study is to determine whether the intervention of delaying cord clamping for 30 to 45 seconds followed by one milking of the cord while simultaneously lowering the VLBW infants below the introitus will result in less bleeding in the brain and fewer infections while in the Neonatal Intensive Care Unit (NICU) and better motor skills at 7 months corrected age. The investigators will attempt to identify the mechanisms of effect through measurement of biologic markers.

DETAILED DESCRIPTION:
The current obstetrical practice at birth in the United States is that the umbilical cord of the very low birth weight (VLBW) infant is clamped immediately. When immediate cord clamping occurs, up to 25% of the fetal-placental blood volume may be left in the placenta acutely increasing vulnerability to hypovolemia. Hypovolemia can precipitate a cascade of physiologic events including poor tissue perfusion, ischemia, and initiation of the fetal/neonatal inflammatory response. Intraventricular hemorrhage (IVH) is a major cause of brain injury for preterm infants and is a predictor of poor neurodevelopment outcomes. Late onset sepsis (LOS) is also associated with morbidity and mortality in the NICU and later developmental delay. Of the approximately 57,000 infants born annually at less than 1500 grams, 10% develop cerebral palsy and 25 to 50% show later cognitive and behavioral deficits affecting school performance with higher rates found in males. We propose a trial with a sample of 212 randomized infants to validate our prior findings that delaying the cord clamping lowers the incidence of intraventricular hemorrhage and late onset sepsis, and to identify the mechanisms of effect through the study of biologic markers including measurement of cytokines, circulating stem cells, and red cell volume. Enrolled women in preterm labor will be randomized at birth to the immediate cord clamping group or the delayed clamping group. Assessment of motor outcomes is planned at 7 months corrected age. This study will help to establish a scientific basis for the timing of cord clamping of VLBW infants. The innovation of this study is in the simplicity of delaying cord clamping for 30 to 45 seconds and lowering the VLBW infants at birth. This low-tech change in a clinical practice has the potential to reduce the risk of disease and disability and to improve the neonatal and early childhood outcomes for these most vulnerable preterm infants.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women between 24 and 31.6 weeks gestation at risk of delivery
* Vaginal or cesarean birth

Exclusion Criteria:

* Congenital anomaly
* Multiple gestation
* Intent to withhold or withdraw care
* Severe or multiple maternal illnesses
* Mothers who are institutionalized or psychotic

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2008-02; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Very low birth weight (VLBW) infants in the delayed cord clamping (DCC) group will have less intraventricular hemorrhage (IVH) compared to VLBW infants in the immediate clamped (ICC) group | December, 2012
Very low birth weight infants in the delayed cord clamping group will have less late onset sepsis than those in the immediate clamping group | December 2012

SECONDARY OUTCOMES:
VLBW infants in the DCC group will have better motor function at 7 months corrected age | November 2012

CONTACTS AND LOCATIONS:
Overall Officials: Judith S Mercer, PhD, CNM, Principal Investigator — University of Rhode Island, Brown University
Locations (1):
- Women and Infants Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Background] Mercer JS, Vohr BR, McGrath MM, Padbury JF, Wallach M, Oh W. Delayed cord clamping in very preterm infants reduces the incidence of intraventricular hemorrhage and late-onset sepsis: a randomized, controlled trial. Pediatrics. 2006 Apr;117(4):1235-42. doi: 10.1542/peds.2005-1706. PMID 16585320
- [Derived] Wang M, Mercer JS, Padbury JF. Delayed Cord Clamping in Infants with Suspected Intrauterine Growth Restriction. J Pediatr. 2018 Oct;201:264-268. doi: 10.1016/j.jpeds.2018.05.028. Epub 2018 Jun 25. PMID 29954605
- [Derived] Mercer JS, Erickson-Owens DA, Vohr BR, Tucker RJ, Parker AB, Oh W, Padbury JF. Effects of Placental Transfusion on Neonatal and 18 Month Outcomes in Preterm Infants: A Randomized Controlled Trial. J Pediatr. 2016 Jan;168:50-55.e1. doi: 10.1016/j.jpeds.2015.09.068. Epub 2015 Nov 4. PMID 26547399
- [Derived] Sommers R, Stonestreet BS, Oh W, Laptook A, Yanowitz TD, Raker C, Mercer J. Hemodynamic effects of delayed cord clamping in premature infants. Pediatrics. 2012 Mar;129(3):e667-72. doi: 10.1542/peds.2011-2550. Epub 2012 Feb 13. PMID 22331336